CLINICAL TRIAL: NCT01152658
Title: Double Blind Prospective Randomize Trail of Partial Tear of SSP and Treatment With PRGF
Brief Title: Partial Tear of Supraspinatus (SSP) and Treatment With Plasma Rich in Growth Factors (PRGF)
Acronym: PrgfRC001IL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC10008-2010CTIL
Record Dates: First submitted 2010-04-26; First posted 2010-06-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2012-03

CONDITIONS: Partial Supraspinatus Tear
Keywords: Partial supraspinatus tear; partial tear ssp per echo
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nacl Injection (Placebo Comparator): 1. Blood samples (4 test tubes) will be extracted from control groups and 8 test tubes for the trial group. The blood of the trial group will be centrifuged and the platelet fraction extracted and counted (only 4 test tubes).
  2. NACL0.9% solution will be then injected to the control group in sterile conditions under ultrasound control
  double blind procedure
  .
  Interventions: Other: NACL
- PRGF (Experimental): 1. Blood samples (4 test tubes) will be extracted from control groups and 8 test tubes for the trial group. The blood of the trial group will be centrifuged and the platelet fraction extracted and counted (only 4 test tubes).2. The enriched plasma fraction will be then injected to the trial group in sterile conditions under ultrasound control.
  Interventions: Biological: PRGF

INTERVENTIONS:
Biological: PRGF — enriched plasma fraction will be then injected to the trial group in sterile conditions under ultrasound control in the ssp gap
  Other Names: trial group
  Arms: PRGF
Other: NACL — Nack 0.9 5 will be then injected to the control group group in sterile conditions under ultrasound control
  Other Names: control group
  Arms: Nacl Injection

SUMMARY:
The objective of this clinical trial is to evaluate the impact and symptomatic efficacy of platelets rich plasma (PRP \ PRGF) in the treatment of partial tears of supraspinatus tendon of rotator cuff.

Speed of tendon healing of partial thickness tear of the supraspinatus tendon influenced by local injection of platelets rich plasma

DETAILED DESCRIPTION:
Primary endpoint: evaluate functional changes after treatment with local infection with platelets rich plasma. This functional changes will be evaluate with Constant Score (questionnaire of shoulder function) and clinical examination.

Secondary endpoint: evaluate the healing effect of the platelets rich plasma locally injected on partial tear of SSP tendon. These morphologic changes will be evaluated by echography

Selection and withdrawal of subjects 40 patients with partial tear of supraspinatus tendon diagnosed by echography. INCLUSION CRITERIA Male or female patients aged between 18 and 60 Patients suffering from partial tear of supraspinatus tendon on echography. Patients who are willing to participate in the trial, to come to all scheduled visits and to sign the informed consent forms.

EXCLUSION CRITERIA Patients receiving other methods of treatment to this area, who had concomitant other injury of the Rotator Cuff tendons.

Non cooperative patient with the basic rehab program.

Trial design

1st visit: Enrollment of patient

1. The patient will be given a full verbal and written explanation regarding the trial and treatment. The patient will sign the informed consent form and will be given a serial number.
2. The screening forms will be completed.
3. Demographic data: date of birth, sex, age and complete medical history, height and previous treatments will be recorded.
4. Fill out questionnaire of shoulder function. Constant score. SST ( Simple shoulder test)
5. Clinical examination will be performed. The results will be recorded in the CRF.
6. Radiology studies: RX Shoulder AP+LAT+ SSP OUTLET VIEW (as required in normal examination of RC injury)
7. Each patient will receive a physiotherapy treatment order according to the protocol of each social work

Randomized separation of the patients in two groups: Control group and the trail group. Patients and medical staff do not know to which group they belong. Double blind trial. (Outside the physician in charge of preparing the blood and the principal investigator)

2nd visit: autologous platelet-rich plasma

1. Blood samples (4 test tubes) will be extracted from control groups and 8 test tubes for the trial group. The blood of the trial group will be centrifuged and the platelet fraction extracted and counted (only 4 test tubes).
2. The enriched plasma fraction will be then injected to the trial group in sterile conditions under ultrasound control. The control group will receive NACL0.9% solution under the same conditions.

3rd visit: 1sr trimester control

1. Fill out questionnaire of shoulder function. Constant score. SST ( Simple shoulder test)
2. Clinical examination will be performed. . Constant score The results will be recorded in the CRF
3. Ultrasound shoulder examination

4rd visit: 2nd trimester control

1. Fill out questionnaire of shoulder function. Constant score. SST (simple shoulder test)
2. Clinical examination will be performed. . Constant score The results will be recorded in the CRF
3. Ultrasound shoulder examination

5th visit: 3rd trimester control

1. Fill out questionnaire of shoulder function. Constant score. STT ( simple shoulder test)
2. Clinical examination will be performed. . Constant score The results will be recorded in the CRF
3. Ultrasound shoulder examination

6th visit: 4th trimester control

1. Fill out questionnaire of shoulder function. Constant score. SST ( simple shoulder test)
2. Clinical examination will be performed. . Constant score The results will be recorded in the CRF
3. Ultrasound shoulder examination
4. End of trial

After one year if treatment if PRGF is proved to be significantly effective on the result of the trail the medical staff is committed to provide treatment, with rich plasma to control patients at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 60
* Patients suffering from partial tear of supraspinatus tendon on echography.
* Patients who are willing to participate in the trial, to come to all scheduled visits and to sign the informed consent forms.

Exclusion Criteria:

* Patients receiving other methods of treatment to this area, who had concomitant other injury of the Rotator Cuff tendons.
* Non cooperative patient with the basic rehab program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
partial tear of supraspinatus tendon | one year

SECONDARY OUTCOMES:
efficacy of platelets rich plasma (PRP \ PRGF) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Palmanovich, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Orthopedic Department - Meir Medical Center, Kfar Saba, Israel